CLINICAL TRIAL: NCT02179671
Title: A Phase IIa, Open-Label, Multi-Center, Multi-Cohort, Immune-Modulated Study of Selected Small Molecules (Gefitinib, AZD9291, or Selumetinib + Docetaxel) or a 1st Immune-Mediated Therapy (IMT; Tremelimumab) With a Sequential Switch to a 2nd IMT (MEDI4736) in Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer (Stage IIIB-IV)
Brief Title: Immune-Modulated Study of Selected Small Molecules (Gefitinib, AZD9291, or Selumetinib + Docetaxel) or a 1st Immune-Mediated Therapy (IMT; Tremelimumab) With a Sequential Switch to a 2nd IMT (MEDI4736) in Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00011
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Locally Advanced or Metastatic Non-Small-Cell Lung Cancer (Stage IIIB-IV)
Keywords: Lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gefitinib; osimertinib; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gefitinib with a Seq. Switch to a MEDI4736 (Experimental): Gefitinib once daily followed by MEDI4736
  Interventions: Drug: Gefitinib
- AZD9291 with a Seq. Switch to a MEDI4736 (Experimental): AZD9291 once daily followed by MEDI4736
  Interventions: Drug: AZD9291
- Selumetinib+Docetaxel with a Seq. Switch to a MEDI4736 (Experimental): Selumetinib twice daily + docetaxel, followed by MEDI4736
  Interventions: Drug: Selumetinib+Docetaxel
- Tremelimumab with a Seq. Switch to a MEDI4736 (Experimental): Tremelimumab every 4 weeks followed by MEDI4736
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Gefitinib — Gefitinib once daily followed by MEDI4736
  Arms: Gefitinib with a Seq. Switch to a MEDI4736
Drug: AZD9291 — AZD9291 once daily followed by MEDI4736
  Arms: AZD9291 with a Seq. Switch to a MEDI4736
Drug: Selumetinib+Docetaxel — Selumetinib twice daily + docetaxel, followed by MEDI4736
  Arms: Selumetinib+Docetaxel with a Seq. Switch to a MEDI4736
Drug: Tremelimumab — Tremelimumab every 4 weeks followed by MEDI4736
  Arms: Tremelimumab with a Seq. Switch to a MEDI4736

SUMMARY:
Primary objective: To assess the efficacy of various sequences of either a small molecule or an IMT (IMT-A) followed by a IMT-B (MEDI4736) .

DETAILED DESCRIPTION:
This is a multi-arm, multi-cohort, Phase IIa, open-label study of selected small molecules (gefitinib, AZD9291, or selumetinib + docetaxel) or 1st IMT (hereafter referred to as IMT-A; tremelimumab) followed by sequential switch to a 2nd IMT (hereafter referred to as IMT-B; MEDI4736) in locally advanced or metastatic NSCLC (Stage IIIB-IV). Patients will be enrolled concurrently into multiple cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Provision of archived tumor tissue sample and mandatory tissue biopsy
* Patients must have either histologically or cytologically documented NSCLC who present with locally advanced or metastatic stage IIIB-IV disease
* Life expectancy ≥12 weeks
* Patients must have measurable disease and at least 1 lesion not previously irradiated
* World Health Organization (WHO) performance status of 0 or 1

Exclusion Criteria:

* Mixed small cell and NSCLC histology
* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2016-06-11 (Actual); Study Completion 2016-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Principal Investigator — International Coordinating Investigator
Locations (10):
- United States (10):
  - Research Site, Goodyear, Arizona
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Augusta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Ashland, Kentucky
  - Research Site, St Louis, Missouri
  - Research Site, Mineola, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 study centers in United States. The first subject was enrolled on 25 July 2014.
Pre-assignment Details: Due to the small numbers of patients treated in Cohorts A through C (gefitinib, AZD9291, or selumetinib + docetaxel), statistical analyses were only done and summary tables prepared for the 28 patients randomised to Cohort D (tremelimumab, either 1-cycle or 2-cycles).
Groups:
- Gefitinib With a Seq. Switch to a MEDI4736: Gefitinib once daily followed by MEDI4736 - analyses not done due to low n
- AZD9291 With a Seq. Switch to a MEDI4736: The 1 patient in the AZD9291 cohort was not dosed and no baseline data were recorded in the database.
- Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736: Selumetinib twice daily + docetaxel, followed by MEDI4736 - analyses not done due to low n
- Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736: Tremelimumab every 4 weeks (1 cycle) followed by MEDI4736
- Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736: Tremelimumab every 4 weeks (2 cycles) followed by MEDI4736
Period: Overall Study
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Started | 1 | 1 | 2 | 14 | 14
Completed | 0 | 0 | 1 | 1 | 1
Not Completed | 1 | 1 | 1 | 13 | 13

BASELINE CHARACTERISTICS:
Population: The 1 patient in the AZD9291 cohort was not dosed and no baseline data were recorded in the database. Because the AZD9291 with a Seq. Switch to a MEDI4736 arm had no data recorded during the study, this arm is not included in the reporting of adverse events.
Groups:
- Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736: TREMELIMUMAB 10MG/KG Q4W 8WEEKS/MEDI4736 10MG/KG Q2W 12MONTHS
- Total: Total of all reporting groups
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Total
Number analyzed (Participants) | 1 | 2 | 14 | 13 | 0 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.0 (0) | 65.0 (12.73) | 57.8 (12.05) | 64.3 (7.85) |  | 61.8 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 6 | 4 |  | 11
  Male | 1 | 1 | 8 | 9 |  | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 2 | 12 | 11 |  | 23
  Black or African American | 0 | 0 | 2 | 2 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Complete Response (CR) Rate
Description: To assess the efficacy of various sequences. CR (per RECIST 1.1 as assessed by the local/site Investigator) is defined as the disappearance of all target and non-target lesions. Confirmed complete response rate (CR rate) is defined as the number (%) of patients with a confirmed overall response of CR and was based on the evaluable analysis set.
Time Frame: Up to 2 years
Population: Per the analysis plan, efficacy would not be analyzed for treatment groups that did not have a sufficient number of enrolled patients.
Measure: Number (80% Confidence Interval); unit: patients (%)
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 7
patients (%) |  |  |  | 0 [NA to NA] — CR=0 | 0 [NA to NA] — CR=0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: To further assess the efficacy of various sequences. Objective response rate (ORR; per RECIST 1.1 as assessed by the site Investigator) is defined as the number (%) of patients with a confirmed overall response of CR or PR and was based on the evaluable analysis set. Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: patients (%)
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 7
patients (%) |  |  |  | 11.1 [1.2 to 36.8] | 0 [NA to NA] — ORR=0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (per RECIST 1.1 as assessed by Investigator) is defined as the date of 1st dose of MEDI4736 until the date of objective disease progression or death. Progression of disease (PD) At least a 20% increase in the sum of diameters of TLs, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 7
patients |  |  |  | 1 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR; per RECIST 1.1 as assessed by the site Investigator) will be defined as the time from the date of 1st documented response (which is subsequently confirmed) until the 1st date of documented progression or death in the absence of disease progression.
Time Frame: Within 12 months
Population: Per the analysis plan, efficacy would not be analyzed for treatment groups that did not have a sufficient number of enrolled patients. Response was observed for 1 patient in the Tremelimumab 1-cycle arm for up to and including 6 months.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
Months |  |  |  | NA — Median was not reached. |

5. Secondary Outcome: Overall Survival
Description: To assess the efficacy of various sequences. In survival follow up at data cut off.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 7
patients |  |  |  | 0 | 0

ADVERSE EVENTS:
Groups:
- AZD9291 With a Seq. Switch to MEDI4736: The 1 patient in the AZD9291 cohort was not dosed and no data were recorded in the database.
Arm/Group | Gefitinib With a Seq. Switch to a MEDI4736 | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 | AZD9291 With a Seq. Switch to MEDI4736 | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/0 | 5/14 | 8/13
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 0/0 | 13/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib With a Seq. Switch to a MEDI4736 (N=1) | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 (N=2) | AZD9291 With a Seq. Switch to MEDI4736 (N=0) | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 (N=14) | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736 (N=13)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib With a Seq. Switch to a MEDI4736 (N=1) | Selumetinib+Docetaxel With a Seq. Switch to a MEDI4736 (N=2) | AZD9291 With a Seq. Switch to MEDI4736 (N=0) | Tremelimumab (1 Cycle) With a Seq. Switch to a MEDI4736 (N=14) | Tremelimumab (2 Cycles) With a Seq. Switch to MEDI4736 (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 | 2 (2) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 2 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 | 3 (3) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 | 6 (10) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 4 (5) | 4 (7)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 2 (2) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 | 4 (6) | 3 (5)
Chills (General disorders) | 0 (0) | 1 (1) | 0 | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 | 6 (6) | 5 (5)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 | 2 (3) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 5 (6)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 | 3 (4) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 | 0 (0) | 4 (4)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 2 (3) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 | 3 (5) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 | 2 (2) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 5 (5) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 2 (2) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 | 3 (5) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 2 (3) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 1 (1) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 | 1 (1) | 1 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No